CLINICAL TRIAL: NCT04559763
Title: SpO2 Accuracy Validation of the OxySoft Sensor Via Reference CO-Oximetry, During Motion and Non-Motion Conditions in Healthy, Well-Perfused Subjects
Brief Title: SpO2 Accuracy Validation of the OxySoft Sensor Via Reference CO-Oximetry Motion Study
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20006OXYVMT
Record Dates: First submitted 2020-08-14; First posted 2020-09-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hypoxia; Desaturation of Blood
Keywords: Oxygen Saturation; Invasive Controlled Desaturation
MeSH Terms: conditions — Hypoxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers
  Interventions: Device: Non-Invasive Controlled Hypoxia; Other: Introduction of Motion conditions: tapping or rubbing

INTERVENTIONS:
Device: Non-Invasive Controlled Hypoxia — Following arterial cannulation, hypoxia is induced by reducing the percent of inspired oxygen the subject breathes while simultaneous measurements are recorded from the test pulse oximeters and arterial blood samples are collected at targeted levels of saturation.
  Other Names: Desaturation; Blood Sampling
Other: Introduction of Motion conditions: tapping or rubbing — Standard motions include tapping or rubbing at periodic intervals with amplitudes of 1-2 cm and 1-4 Hz with a random variation in frequency will occur at each plateau. Each plateau will have both an interval of tapping and rubbing. Signals are recorded by a validated, computerized data acquisition system (CAS). The device values are sampled once per second and averaged over the time taken to draw the blood sample, taking into account circulation time delays and differences in device response times

SUMMARY:
SpO2 (oxygen saturation) and pulse rate accuracy of pulse oximetry equipment, OxySoft Sensor/N-600x and OxySoft Sensor/N-395, continuous measure of arterial oxygen saturation during hypoxic state throughout motion and non-motion conditions under one system configuration.

The purpose of this Non-Randomized, Prospective,Observational study is to conduct a hypoxia study to directly compare a prototype OxySoft pulse oximeter system to arterial oxygen saturation.

DETAILED DESCRIPTION:
The study utilizes a single-site, physiology laboratory for non-randomized, prospective, interventional studies. The goal is to enroll a range of twelve (12) to sixteen (16) healthy adult volunteers. Subjects may be of any race,ranging in pigmentation from light to dark to meet the study design requirements.

The general purpose of Invasive Controlled Desaturation Studies during motion is to validate the SpO2and pulse rate accuracy in comparison to reference-standard measurements of blood SaO2 by a CO-oximeter during motion conditions. This is achieved through paired observations of SpO2 and SaO2values over the specified SpO2 accuracy range of 70 % to 100 % SaO2 of the prototype pulse oximeter on a group of healthy adult volunteers. The fraction of inspired oxygen (FiO2) delivered to test subjects is varied to achieve a series of targeted steady-state saturation periods. Arterial blood samples are periodically taken from an indwelling arterial catheter for use in the comparison.

Pulse rate accuracy will be evaluated during the same data collection period as SpO2. Pulse rate will be compared to reference ECG heart rate.In the unlikely event that the ECG monitor malfunctions, the Pulse rate reference may be taken using the average pulse rate value from the transfer standard pulse oximeters. This study is designed to support an FDA submission for pulse rate and saturation accuracy in a diverse subject population during motion conditions over a specified saturation range for the Oxysoft pulse oximetry system.

The FDA Guidance Document for Pulse Oximeters and ISO 80601-2-61 define the accepted guideline for evaluation and documenting the SpO2 accuracy in humans. The OxySoft sensor is not FDA approved for the intended study population, healthy adults. To support the development of Nellcor pulse oximeter systems, data is required to test the performance of the sensors with pulse oximetry systems in the adult patient population. In order to accurately validate sensors, manipulation of oxygen and nitrogen levels through the administration of oxygen and nitrogen gas will occur. Measurements of SpO2and pulse rate accuracy in comparison to reference-standard measurements of blood SaO2 by a CO-oximeter during motion and non-motion conditions will be taken and analyzed to support development of Nellcor technology and support FDA submission.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand and provide written informed consent
2. Adult subjects 18 to 50 years of age.
3. Subject must be willing and able to comply with study procedures and duration.
4. Subject is a non-smoker or who has not smoked within 2 days prior to the study.
5. Male or female of any race.
6. Cleared same day Health Assessment form and health screening.
7. Subject demographics include a range of skin pigmentations, including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger.
8. Successful Perfusion Index Ulnar/Ulnar+Radial Ratio test showing adequate collateral blood flow.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Subject is considered as being morbidly obese (defined as BMI >39.5)
2. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized.)
3. Females of childbearing potential, who are pregnant, who are trying to get pregnant or who have a urine test positive for pregnancy on the day of the study
4. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
5. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
6. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
7. Subjects with known respiratory conditions such as:

   1. uncontrolled / severe asthma,
   2. flu,
   3. pneumonia / bronchitis,
   4. shortness of breath / respiratory distress,
   5. unresolved respiratory or lung surgery,
   6. emphysema, COPD, lung disease
8. Subjects with known heart or cardiovascular conditions such as:

   1. Hypertension: systolic >140mmHg, or Diastolic >90mmHg on 3 consecutive readings.
   2. have had cardiovascular surgery
   3. Chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or
   5. with respiratory sinus arrhythmia
   6. previous heart attack
   7. blocked artery
   8. unexplained shortness of breath
   9. congestive heart failure (CHF)
   10. history of stroke
   11. transient ischemic attack
   12. carotid artery disease
   13. myocardial ischemia
   14. myocardial infarction
   15. cardiomyopathy
9. Self-reported health conditions as identified in the Health Assessment Form

   1. diabetes,
   2. uncontrolled thyroid disease,
   3. kidney disease / chronic renal impairment,
   4. history of seizures (except childhood febrile seizures),
   5. epilepsy,
   6. history of unexplained syncope,
   7. recent history of frequent migraine headaches,
   8. recent symptomatic head injury, within the last 2 months
   9. Subjects with known clotting disorders
   10. history of bleeding disorders or personal history of prolonged bleeding from injury
   11. history of blood clots
   12. hemophilia
   13. current use of blood thinner: prescription or daily use of aspirin
   14. Subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
   15. Subjects with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
   16. Arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site. left or right)
   17. History of clinically significant complications from previous arterial cannulation.
   18. A radial artery with ten or more arterial cannulations right or left, excludes that site.
   19. Unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits.
   20. Other known health condition, should be considered upon disclosure in Health Assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be a minimum of twelve subjects, ranging in pigmentation from light to dark to skin tones including subjects with deep pigmentation and the subject selection will be an equitable distribution of males and females.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
To investigate performance of the OxySoft device by measuring oxygen saturation accuracy during motion and non-motion conditions | October 2020
  The primary objective of the study is to investigate the efficacy and performance of the OxySoft device by measuring oxygen saturation accuracy in a diverse subject population during motion and non-motion conditions and over a specified saturation range.
  The acceptance criteria for SpO2, on the non-motion hand, across the saturation range of 70-100% when paired with the N-395:
  SpO2 OxySoft Sensor/N-395 ± 3% (Arms)
  The acceptance criteria for SpO2 during motion conditions, on the motion hand, across the saturation range of 70-100% when paired with the N-600x:
  SpO2 OxySoft Sensor/N-600x ± 3% (Arms)
To investigate efficacy and performance of OxySoft device by measuring pulse rate accuracy during motion and non-motion conditions | October 2020
  The secondary objective of the study is to investigate the efficacy and performance of the OxySoft device by measuring pulse rate accuracy in a diverse subject population during motion and non-motion conditions and over a specified saturation range.
  The acceptance criteria for pulse rate during motion conditions, on the motion hand, across the saturation range of 70-100% when paired with the N-600x:
  PR OxySoft Sensor/N-600x ≤ 5 BPM

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be analyzed and outlined in final study report. Individual participant data will only be made available to the participant and or participant primary care physician as applicable.